CLINICAL TRIAL: NCT04572776
Title: A Multicenter, Randomized, 2-Arm, Phase 3 Study to Assess the Efficacy and Safety of a Single Epidural Administration of Resiniferatoxin Versus Standard of Care (SoC) for the Treatment of Intractable Pain Associated With Cancer
Brief Title: Phase 3 Study to Assess Resiniferatoxin vs Standard of Care for the Treatment of Intractable Cancer Pain
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: To be replaced by a different protocol
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STI-RTX-300x
Record Dates: First submitted 2020-09-29; First posted 2020-10-01 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Pain, Intractable; Pain Cancer
Keywords: pain; cancer pain; intractable pain; RTX; resiniferatoxin
MeSH Terms: conditions — Pain, Intractable; Cancer Pain; Pain | interventions — resiniferatoxin; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Follow-up visit examinations will be performed by a blinded outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resiniferatoxin (Experimental): Single dose of Resiniferatoxin (25 mcg in 3 mL) injected epidurally
  Interventions: Drug: Resiniferatoxin
- Standard of Care (Active Comparator): Standard of care treatment as determined by the investigator
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Resiniferatoxin — Resiniferatoxin is a TRPV-1 agonist which works by specifically ablating nociceptive nerve fibers.
  Other Names: RTX
  Arms: Resiniferatoxin
Other: Standard of Care — Standard of care for intractable pain with the exception of intra-thecal pump placement as determined by the investigator.
  Other Names: SOC
  Arms: Standard of Care

SUMMARY:
This is a Phase 3 study to assess the safety and efficacy of a single epidural administration of Resiniferatoxin versus standard of care for the treatment of intractable pain associated with cancer.

DETAILED DESCRIPTION:
This study is a multicenter, randomized Phase 3 study to assess the safety and efficacy of a single epidural administration of Resiniferatoxin versus standard of care (SOC) for the treatment of intractable pain associated with cancer. Subjects will be followed for 12 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed clinical diagnosis of advanced cancer or metastasis.
* Pain in the target area (lower thoracic or chest level down to lower extremities) most likely attributed to cancer as per Investigator.
* Pain severity at the target area is moderate-to-severe, defined as worst pain ≥6 on the NPRS during screening (average of the 3 days prior to Day 1), despite available pain therapy or analgesia. Subjects with multiple sites of pain are eligible as long as the intensity of pain at the intended target location for treatment fulfills the score of ≥6 and can be differentiated from other areas.
* Must report NPRS scores in the daily diary for at least 3 days prior to Day 1.
* Must be at least 18 years of age or older at Screening.
* Subject has reasonable expectation that they will be able to complete the study (through at least the week 4 visit).
* Life expectancy of at least 6 months at screening
* Minimum Karnofsky score of 50 at screening
* Sexually active female participants of childbearing potential must be willing to use an effective method of contraceptive method to avoid pregnancy
* Must have provided written informed consent which includes signing the institutional review board approved consent form prior to participating in any study related activity.
* Must be willing and capable of understanding and cooperating with the requirements of the study, including the ability to perform/undergo all required assessments for the duration of the study.
* Must be able to understand, and complete study related forms and adequately communicate with the investigator and/or site staff.

Exclusion Criteria:

* Undergoing or have plans to undergo changes to current cancer treatment from 7 days prior to Day 1 to 4 weeks after Day 1. Continuation of existing anti-cancer therapy without any planned change in dose or regimen is permitted. Participants may receive new cancer therapy 4 weeks after Day 1 including investigational agents in another clinical trial while participating in this study. If participating in another trial, it is requested that the subject agree to continue clinic visits and completion of patient diaries in this trial.
* Participants with leptomeningeal metastases in the lumbar area.
* Level of intended epidural injection is in the site of prior lumbar spine surgical procedures, such as posterior spinal fusions, that could impair the ability to perform the injection, as assessed by the Investigator.
* Evidence of increased intracranial pressure as determined by symptoms, history, physical examination, and/or magnetic resonance imaging (MRI).
* Patients with an intra-thecal pump implanted within 2 weeks of the baseline visit will be excluded. Pump placement during the study will not be permitted for 4 weeks after the study drug is administered; and existing pump medications cannot be changed during that same initial 4 week period.
* Has evidence of a non-correctable coagulopathy or hemostasis problem at Screening (V1) or Baseline (V2) as defined by:
* Prothrombin Time/International Normalized Ratio ≥1.3 times upper limit of normal (ULN) range with blood drawn within 1 week of the planned injection.
* Partial thromboplastin time ≥1.5times upper limit of normal (ULN) with blood drawn within 1 week of the planned injection.
* Platelet count <75,000 cells/mm3 with blood drawn within 1 week of the planned injection. Participants must stop any anticoagulant (e.g., warfarin) or antiplatelet (e.g., aspirin) before and during IP administration according to acceptable medical guidelines. Participants with abnormal PT or PTT at Screening, but whose PT or PTT is expected to normalize once anticoagulation is held, are eligible as long as the PT or PTT has normalized prior to the planned injection.
* Participants with a total neutrophil count <750 cells/mm3 at Screening (V1) or Baseline (V2).
* Is febrile or has other evidence of an infection within 24 hours of the planned injection.
* Has an allergy or hypersensitivity to capsaicin, or radiographic contrast agents used in diagnostic imaging studies.
* Female participants who are pregnant at Screening (V1) or Day 1 (V2), are planning on becoming pregnant, or are currently breastfeeding.
* Participants with any medical condition that, in the Investigator's opinion, could adversely impact study participation or safety, the conduct of the study, or interfere with the pain assessments.
* Participants with additional loci of pain above the midthoracic level or other pain disorder due to noncancer etiology at Screening (V1), unless both the investigator and the subject are clearly able to distinguish this pain from the target pain due to cancer.
* Non-study related minor surgical procedure ≤2 days or major surgical procedure ≤7 days prior to the Screening Visit. In all cases, the subject must be sufficiently recovered and stable prior to IP administration on D1.
* Participants who have not recovered from any toxicities from previous chemotherapy, hormone therapy, immunotherapy, or radiotherapies that are Grade 3 or higher by CTCAE. Participants are eligible if the toxicities are Grade 2 or less, as long as all other inclusion/exclusion criteria are fulfilled.
* Arterial thrombi (including stroke), myocardial infarction, admission for unstable angina, within 3 months prior to Screening (V1).
* Evidence or history of bleeding disorder, i.e., any hemorrhage or bleeding event of CTCAE >Grade 2 within 4 weeks prior to D1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in worst pain as assessed using the Numeric Pain Rating Scale (NPRS) | Baseline to Week 4
  Change from baseline to Week 4 in the intensity of worst pain over the previous 24 hours in the area targeted for treatment as measured by the 11-point NPRS (0-10 where 0 is no pain and 10 is worst pain imaginable)

SECONDARY OUTCOMES:
Change in worst pain as assessed using the NPRS | Baseline to Weeks 8 and 12
  Change from baseline to Weeks 8 and 12 in the intensity of worst pain over the previous 24 hours in the area targeted for treatment as measured by the 11-point NPRS (0-10 where 0 is no pain and 10 is worst pain imaginable)
Change in area under the curve (AUC) of worst pain as assessed using the NPRS | Baseline through Week 4
  AUC calculated on change from baseline through Week 4 in worst pain in the target pain location over the previous 24 hours, using the NPRS (0-10)
Incidence and severity of adverse events (AEs) | Baseline through Week 12
  Incidence and severity of AEs assessed using the Common Terminology Criteria for Adverse Events (CTCAE) criteria
Change in Quality of Life (QOL) as assessed using the modified Brief Pain Inventory-Short Form (BPI-SF) | Baseline to Week 4
  Change in Quality of Life from baseline to week 4 based on total score from the BPI-SF, modified to record the target pain treated with study drug
Duration of response in subjects who experienced ≥20% decrease from baseline in worst pain as assessed using the NPRS | Randomization through Week 12
  Duration of response defined as time from ≥20% decrease from baseline in worst pain score in the target pain location to ≥20% increase from the nadir of the worst pain score
Change in intensity of average pain as assessed using the NPRS | Baseline to Week 4
  Change from baseline to Week 4 in the intensity of average pain over the previous 24 hours in the target pain location as measured by the NPRS (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Luchi, MD, Study Director — Sorrento Therapeutics